CLINICAL TRIAL: NCT06172387
Title: The Efficacy of Intra-arterial Albumin With Endovascular Treatment for Acute Ischemic Stroke : A Randomized, Controlled Pilot Study
Brief Title: Intra-arterial Albumin in Acute Ischemic Stroke After Endovascular Treatment for
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tianjin Huanhu Hospital (Other)
Responsible Party: Principal Investigator, Ming Wei, Chief physician, Tianjin Huanhu Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TJHH-2023-WM121
Record Dates: First submitted 2023-12-07; First posted 2023-12-15 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Acute Ischemic Stroke
Keywords: acute ischemic stroke; albumin; intra-arterial; thrombectomy; neuroprotection
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intra-arterial group (Experimental): 20% human serum albumin (0.6g/kg) solution will be injected into the artery after revascularization in acute ischemic stroke. All participants will receive mechanical thrombectomy and a standard clinical therapy.
  Interventions: Drug: intra-arterial infusion albumin; Other: mechanical thrombectomy and a standard clinical therapy
- sham group (Other): All participants have no intra-arterial albumin.
  Interventions: Other: mechanical thrombectomy and a standard clinical therapy

INTERVENTIONS:
Drug: intra-arterial infusion albumin — The experimental group would inject 20% human blood albumin solution into the responsible blood vessel supply area by catheter artery at a dose of 0.6g/kg. The infusion time is 20-30 minutes. All participant will receive mechanical thrombectomy and a standard clinical therapy.
  Arms: intra-arterial group
Other: mechanical thrombectomy and a standard clinical therapy — mechanical thrombectomy and a standard clinical therapy

SUMMARY:
Stroke is an acute focal injury of the central nervous system caused by cerebral vessels. One in every four people is affected by stroke at different times in life. Globally, stroke is the second leading cause of death and third leading cause of disability in adults. we hypothesized that in patients with acute large vessel occlusive ischemic stroke treated with mechanical thrombectomy, the infusion of 20% human serum albumin solution into the revascularization area can exert a stronger neuroprotective effect.

DETAILED DESCRIPTION:
In the previous period, we have conducted a clinical trial on the safety and feasibility of arterial infusion of 20% human serum albumin solution. The results of the study found that after arterial infusion of 20% human serum albumin solution at a dose of 0.6g/kg to the subject's vascularization area, the subjects did not develop significant complications related to albumin solution. There were no serious adverse events associated with arterial infusion of albumin solution in all subjects. After the evaluation of the Data Safety Monitoring Board, the clinical study was considered to be the next step, which is to initially explore the effectiveness of 0.6g/kg arterial infusion of 20% human serum albumin solution for neuroprotection of subjects.

ELIGIBILITY:
Inclusion Criteria:

1.Male or female, age≥18 and ≤ 80; 2. anterior circulation large vessel occlusion confirmed by CTA, MRA and DSA; 3. baseline National Institute of Health Stroke Scale (NIHSS) score ≥6； 4. Alberta Stroke Program Early CT Score (ASPECTS) 6-10; 5. Stroke symptoms present to femoral artery or brachial artery puncture within 24 hours； 6. occluded vessel reaches eTICI level ≥2b after thrombectomy confirmed by DSA；7. Informed consent obtained;

Exclusion Criteria:

(1) history of congestive heart failure or jugular dilatation, third heart sound, resting tachycardia due to heart failure (>100 beats/min), hepatomegaly and lower limb edema without obvious cause on admission physical examination; (2) hospitalization for acute myocardial infarction within 3 months; (3) symptoms of acute myocardial infarction or admission electrocardiogram; (4) second or third degree heart block or arrhythmia with hemodynamic instability; (5) acute or chronic renal failure (blood creatinine > 2.0 mg/dL); (6) severe anemia (hematocrit<32%); (7) symptoms or CT evidence of subarachnoid hemorrhage; (8) pregnancy; (9) allergy to albumin; (10) admission blood pressure higher than 185/110 mmHg; (11) any chronic lung disease, including chronic obstructive pulmonary disease, bronchiectasis, and other lung diseases that interfere with daily activities; (12) presence of other diseases that may endanger life.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
cerebral infarct volume | 24-48 hours after randomization
  infarct volume is evaluated mainly through brain MRI

SECONDARY OUTCOMES:
modified Rankin Scale score(mRS) | 90 ±10 days after randomization
  the mRS is an ordinal disability score of 7 categories (0=no symptoms to 5=severe disability, and 6=death)
the good prognosis at 90 days assessed by mRS | 90 ±10 days after randomization
  the mRS is an ordinal disability score of 7 categories (0=no symptoms to 5=severe disability, and 6=death)
scores assessed by National Institutes of Health Stroke Scale (NIHSS) | 24 ± 6 hours, 48 ± 12 hours, 7 ± 2 days, 90 ±10 days after randomization
  the NIHSS is a stroke severity score that is composed of 11 items, range from 0 to 42, higher values indicate more severe deficits
change in National Institutes of Health Stroke Scale (NIHSS) score from baseline to 24 hours | from baseline to 24 ± 6 hours
  the NIHSS is a stroke severity score that is composed of 11 items, range from 0 to 42, higher values indicate more severe deficits
improvement of neurologic function after 24 hours | 24 ± 6 hours after randomization
  NIHSS score decreased by more than 4 points or NIHSS score was 0; secondary clinical efficacy endpoint; the NIHSS is a stroke severity score composed of 11 items (range from 0 to 42, higher values indicate more severs deficits)
Barthel index (BI) | 90 ±10 days after randomization
  the BI is an ordinal disability score of 10 categories (range from 0-100, higher values indicate better prognosis)
revascularization on follow-up imaging | 24 (16 to 36) hours
  secondary imaging efficacy endpoint
24-hours neurologic deterioration | 24 ± 6 hours after randomization
  NIHSS score increased by more than 4 points; the NIHSS is a stroke severity score composed of 11 items (range from 0 to 42, higher values indicate more severe deficits); clinical safety endpoint
any intracranial hemorrhage on follow-up imaging | 24 (12 to 36) hours
  imaging safety endpoints; per ECASSIII definition and per Heidelberg bleeding classification
symptomatic intracerebral hemorrhage | 24 (12 to 36) hours
  imaging safety endpoints; deterioration in NIHSS score of ≥4 point within 24 hours;per ECASS III definition and per Heidelberg bleeding classification
Mortality | 90 ± 10 days after randomization
  clinical safety endpoint
Stroke recurrence | 90 ± 10 days after randomization
  clinical safety endpoint
Survival rates | 7 ± 2 days, 90 ± 10 days after randomization
  secondary clinical efficacy endpoint
mRS4-6 | 90 ± 10 days after randomization
  secondary clinical efficacy endpoint;the mRs is an ordinal disability score of 7 categories (0 = no symptoms to 5 = severe disability, and 6 = death)

CONTACTS AND LOCATIONS:
Locations (1):
- Ming wei, Tianjin, China, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided